CLINICAL TRIAL: NCT00506662
Title: The Effect of Insulin Detemir on Glucose Control in Ageing Subjects With Type 2 Diabetes.
Brief Title: Comparison of Insulin Detemir and NPH Insulin Given Once Daily in Ageing Subjects With Type 2 Diabetes
Acronym: 3L
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1808; 2006-006589-41 (EudraCT Number)
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin detemir (Experimental): Individually adjusted dose of insulin detemir once daily
  Interventions: Drug: insulin detemir
- Insulin NPH (Active Comparator): Individually adjusted dose of insulin NPH once daily
  Interventions: Drug: insulin NPH

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target, s.c. (under the skin) injection, once daily
  Arms: Insulin detemir
Drug: insulin NPH — Treat-to-target, s.c. (under the skin) injection, once daily
  Arms: Insulin NPH

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to compare insulin detemir once daily to NPH insulin once daily as measured by blood sugar control in ageing subjects with type 2 diabetes naive to previous insulin therapy.

DETAILED DESCRIPTION:
Novo Nordisk has decided to discontinue the trial as it will not be possible to recruit the required number of patients. The discontinuation is based on an analysis of the significant delay in recruitment of patients which is likely to have a negative impact on the validity of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin naive
* Treatment with oral anti-diabetic drugs (OADs) for at least 3 months and not achieving therapeutic targets
* HbA1c between 8% - 10.5%

Exclusion Criteria:

* Secondary diabetes, MODY (Maturity Onset Diabetes of the Young)
* Previous treatment with insulin (except for short-term treatment with insulin for intercurrent illness as judged by the Investigator)
* Proliferative retinopathy, maculopathy requiring treatment,
* Hypoglycaemia unawareness as judged by the Investigator, recurrent major hypoglycaemia
* End stage liver disease (increased liver enzymes 4 fold), end stage renal disease assessed by MDRD (Modification of Diet in Renal Disease) less than 30 ml/min or dialysed patient, acute heart failure, any acute cardiovascular event or cerebrovascular event less than 6 months
* Acute disease with poor prognosis
* History of alcoholism, drug abuse, or psychiatric disease or personality disorders likely to invalidate voluntary consent or to prevent good compliance with the trial protocol
* Mental incapacity, unwillingness or language barrier precluding adequate understanding or co-operation (patients having a score of less than 15 in a previous MMSE (Mini-Mental State Examination) in the last six months) and any conditions as judged by the investigator
* Legal incapacity or limited legal capacity (patients under guardianship or curatorship)
* Concomitant medication for Alzheimers treatment (Memantine, Anticholinesterasique treatment)
* Participation in another clinical trial less than one month before inclusion in this trial
* Illness requiring repeated hospitalisation
* Known or suspected allergy to the insulin or any compositional component
* Anticipated change or new use in concomitant medication known to interfere with glucose metabolism, such as systemic corticotherapy more than 5 mg/day (prednisone)
* Any other condition that the Investigator feels would interfere with trial participation or evaluation of results
* Terminal illness

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Paris La Défense, France
- Cambridge, United Kingdom

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 57 centres in 2 countries: France (35) and United Kingdom (22)
Pre-assignment Details: Subjects in the trial were patients with type 2 diabetes being treated with oral anti-diabetic drug (OAD) therapy(ies) for at least 3 months prior to the trial and considered to benefit from insulin treatment. The randomisation target for this trial was 286.
Period: Overall Study
Arm/Group | Insulin Detemir | Insulin NPH
Started | 38 | 48
Completed | 21 | 20
Not Completed | 17 | 28
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 2 | 4
Not completed — Trial terminated | 10 | 16
Not completed — Not recorded | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir | Insulin NPH | Total
Number analyzed (Participants) | 38 | 48 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 38 | 48 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (5.5) | 76.1 (4.9) | 76.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 17 | 29 | 46
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (4.6) | 29.8 (5.5) | 29.5 (5.1)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 13.3 (10.3) | 15.2 (9.4) | 14.6 (9.8)
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total haemoglobin] | 9.26 (0.87) | 9.12 (0.78) | 9.19 (0.82)
Weight [Mean (Standard Deviation); unit: kg] | 77.4 (15.9) | 80.4 (16.4) | 79.0 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) at Month 7
Time Frame: week 0, month 7
Population: Due to the recruitment issue, the trial has been prematurely interrupted and the final number of patients does not allow any efficacy analysis.
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) at Month 4
Time Frame: week 0, month 4
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Mean Fasting Plasma Glucose (FPG) at Month 7
Time Frame: week 0, month 7
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Mean Fasting Plasma Glucose (FPG) at Month 4
Time Frame: week 0, month 4
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Mean Pre-lunch Plasma Glucose at Month 7
Time Frame: week 0, month 7
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Mean Pre-lunch Plasma Glucose at Month 4
Time Frame: week 0, month 4
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Mean Pre-dinner Plasma Glucose at Month 7
Time Frame: week 0, month 7
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Mean Pre-dinner Plasma Glucose at Month 4
Time Frame: week 0, month 4
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Body Weight at Month 7
Time Frame: week 0, month 7
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Body Weight at Month 4
Time Frame: week 0, month 4
Population: as for outcome 1
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Mean Number of Total Hypoglycaemic Episodes, Month 1
Description: Mean number of total hypoglycaemic episodes per patient expressed as rate per week by visit. Rate per week is calculated by dividing the number of episodes for each patient by the number of weeks in the period.
Time Frame: weeks -2-0, month 1
Population: The safety analysis set is all patients who had been exposed to at least one dose of the trial product, and had hypoglycaemia data available at both endpoints.
Measure: Mean (Standard Deviation); unit: episodes per week by visit
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 38 | 48
episodes per week by visit
  Screening (week -2 to week 0) | 0.039 (0.179) | 0.073 (0.372)
  Month 1 (weeks 1-4) | 0.026 (0.097) | 0.120 (0.282)
  Difference (month 1-screening) | -0.013 (0.209) | 0.047 (0.446)

12. Secondary Outcome: Mean Number of Total Hypoglycaemic Episodes, Months 2-4
Description: as for outcome 11
Time Frame: weeks -2-0, months 2-4
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: episodes per week by visit
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 38 | 46
episodes per week by visit
  Screening (week -2 to week 0) | 0.039 (0.179) | 0.076 (0.380)
  Months 2-4 (weeks 5-16) | 0.015 (0.051) | 0.072 (0.167)
  Difference (months 2-4 - screening) | -0.024 (0.177) | -0.004 (0.394)

13. Secondary Outcome: Mean Number of Total Hypoglycaemic Episodes, Months 5-7
Description: as for outcome 11
Time Frame: weeks -2-0, months 5-7
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: episodes per week by visit
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 38 | 43
episodes per week by visit
  Screening (week -2 to week 0) | 0.039 (0.179) | 0.058 (0.381)
  Months 5-7 (weeks 17-28) | 0.018 (0.078) | 0.041 (0.099)
  Difference (months 5-7 - screening) | -0.022 (0.131) | -0.017 (0.400)

ADVERSE EVENTS:
Time Frame: The adverse events were collected from July 2007 to December 2008.
Description: The safety analysis set is all patients who had been exposed to at least one dose of the trial products.
Arm/Group | Insulin Detemir | Insulin NPH
Serious Adverse Events (participants affected / at risk) | 2/38 | 8/48
Other Adverse Events (participants affected / at risk) | 13/38 | 11/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=38) | Insulin NPH (N=48)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Campylobacter intestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=38) | Insulin NPH (N=48)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 4 (6)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (4) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Trial terminated prematurely due to low recruitment, and thus it was not possible to assess efficacy in this trial due to the small number of patients in each treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Steering Committee has the right to publish the entire results of the trial. Any such scientific paper, presentation, communication, or other information concerning the investigation described in this protocol, must be approved by the Steering Committee, and copies submitted in writing to Novo Nordisk prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.